CLINICAL TRIAL: NCT00705770
Title: A Multi-Dose Study With a Treatment for Open-Angle Glaucoma
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Change in study design
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-07-58
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2008-07

CONDITIONS: Open-Angle Glaucoma
Keywords: Open-Angle Glaucoma; Intraocular Pressure; Anecortave Acetate
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — anecortave acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Placebo treatment with vehicle
  Interventions: Drug: Placebo
- 2 (Experimental): Low dose of study medication
  Interventions: Drug: Anecortave Acetate
- 3 (Experimental): Middle dose of study medication
  Interventions: Drug: Anecortave Acetate
- 4 (Experimental): High dose of study medication
  Interventions: Drug: Anecortave Acetate

INTERVENTIONS:
Drug: Anecortave Acetate — Low dose
  Sustained release depot suspension
  Arms: 2
Drug: Anecortave Acetate — Middle dose
  Sustained release depot suspension
  Arms: 3
Drug: Anecortave Acetate — High dose
  Sustained release depot suspension
  Arms: 4
Drug: Placebo — Placebo treatment with vehicle
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether Anecortave Acetate is effective for lowering intraocular pressure caused by open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old with a clinical diagnosis of Open-Angle Glaucoma for at least 6 months and currently treated with a monotherapy hypotensive medication

Exclusion Criteria:

* Prior angle surgery in the study eye, severe visual field loss in either eye, and any other form of glaucoma besides open-angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Mean Intraocular Pressure | 6 months

SECONDARY OUTCOMES:
Percent of patients with therapeutic benefit, number and percent of treatment failure and time to treatment failure | 6 months